CLINICAL TRIAL: NCT00635687
Title: Can Liver Stiffness Values Predict Early Rebleeding in Variceal Rupture
Brief Title: Transient Elastography and Variceal Bleeding
Acronym: PROME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006/102/HP
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Bleeding
Keywords: variceal bleeding; transient elastography
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibroscan (Experimental)
  Interventions: Device: Fibroscan

INTERVENTIONS:
Device: Fibroscan — transient elastography measure - Liver stiffness

SUMMARY:
Transient elastography is a new non-invasive rapid and reproducible method, allowing evaluating liver fibrosis by measurement of liver stiffness.

The aim of our study is to evaluate if the liver stiffness can predict the recurrence of upper variceal bleeding in cirrhotic patients hospitalized for variceal rupture.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed
* Social security affiliation
* Variceal bleeding with hematemesis or melena within 24 hours of inclusion
* Age > 18 years
* Scheduled to undergo endoscopy within 24 hours of hospital admission

Exclusion Criteria:

* Hepatocarcinoma
* Upper Gastro Intestinal bleeding for other causes than variceal bleeding
* Concomitant disease with a life expectancy of less than 45 days
* Rebleeding within 24 hours after first endoscopy
* Technical failure of transient elastography

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-03; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Bleeding recurrence rate | J45 post first hemorrage

CONTACTS AND LOCATIONS:
Overall Officials: Sophie HERVE, MD, Principal Investigator — University Hospital, Rouen
Locations (4):
- France (4):
  - UH Amiens, Amiens
  - UH Caen, Caen
  - UH Lille, Lille
  - Rouen University Hospital, Rouen